CLINICAL TRIAL: NCT05270421
Title: Effect of Furosemide on Outcome of Extracorporeal Shock Wave Lithotripsy for Renal and Ureteral Calculi; a Randomized, Triple-blinded, Controlled Trial
Brief Title: Effect of Furosemide on ESWL Outcomes for Renal and Ureteral Calculi
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyed Hossein Hosseini, Principal Investigator, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21179-01-01-98
Record Dates: First submitted 2022-02-12; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Urolithiasis; Nephrolithiasis; Urinary Calculi; Ureterolithiasis
Keywords: Urolithiasis; Nephrolithiasis; ESWL
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis; Urinary Calculi; Ureterolithiasis | interventions — Furosemide

STUDY DESIGN:
Intervention Model Description: 500 patients will be randomly and equally divided into the intervention and control groups.
Who Masked: Participant, Investigator
Masking Description: Using block randomization, the patients are randomly assigned to one of two groups by a statistician outside of the research group. The codes for each group remain unknown to the researchers until after statistical analysis, with only the nurse and physician in charge of delivering the therapy and monitoring the patients being made aware.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): 40 mg of furosemide IV + IV midazolam + 1000 ml of normal saline 30 minutes before ESWL
  + Standard ESWL
  Interventions: Drug: Furosemide 40 mg; Other: Conventional Treatment
- Control Group (Active Comparator): IV midazolam + 1000 ml of normal saline 30 minutes before ESWL
  + Standard ESWL
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Drug: Furosemide 40 mg — Standard ESWL + Furosemide 40 mg
  Arms: Intervention Group
Other: Conventional Treatment — Standard ESWL

SUMMARY:
The minimally-invasive extracorporeal shockwave lithotripsy (ESWL) procedure is generally considered the best first-line treatment option for most adults and children with nephrolithiasis, especially when the calculi are smaller than 2 cm in size. Despite some promising results, few clinical trials have assessed the impact of furosemide on the outcome of ESWL. This study seeks to determine the effect of furosemide on ESWL outcomes when treating renal and ureteral calculi, hypothesizing that it will result in better outcomes for patients.

The present double-blind, randomized clinical trial includes 500 adults aged 18-60 years referring to the ESWL Clinic of Shahid Faghihi Hospital. Using block randomization, the patients are randomly assigned to one of two groups. All patients are to receive sedation with intravenous midazolam and 1000 ml of normal saline 30 minutes before ESWL. The only difference between the groups is that in the furosemide group, 40 mg of furosemide is added to the normal saline in the drug preparation room before administration. All patients are kept under heart monitoring and pulse oximetry until recovery. Pain will be checked for all participants via a telephone interview 24 hours later. The outcomes and possible side effects of ESWL will be evaluated for all patients after two and twelve weeks.

DETAILED DESCRIPTION:
The present study takes the form of a double-blind, randomized clinical trial. The study conforms to the principles stated in the Declaration of Helsinki. Written informed consent is obtained from all subjects prior to enrolment. All participants are made aware of the study protocol and can withdraw from the study at any point. Given that furosemide does not adversely affect patients who do not have cardiovascular or renal diseases, no complications are predicted. The trial is pending registration with clinicaltrials.gov. This protocol was conceived following the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) guidelines.

By taking into account an alpha error of 0.05 and a test power of 80%, the number of subjects in each group was calculated at 232. Considering a dropout rate of 10%, 250 subjects are to be included in each group.

Using block randomization, the patients are randomly assigned to one of two groups by a statistician outside of the research group. The codes for each group remain unknown to the researchers until after statistical analysis, with only the nurse and physician in charge of delivering the therapy and monitoring the patients being made aware.

All patients are to receive sedation with intravenous midazolam and 1000 ml of normal saline 30 minutes before ESWL, which is to be performed in the standard manner. The only difference between the groups is that in the furosemide group, 40 mg of furosemide is added to the normal saline in the drug preparation room before administration. All patients are kept under heart monitoring and pulse oximetry until recovery. Given that furosemide may theoretically cause pain secondary to hydronephrosis, pain will be checked for all participants via a telephone interview 24 hours later using a visual analog scale (VAS) of 0 to 10.

The outcomes and possible side effects of ESWL are evaluated for all patients after two and twelve weeks. A KUB X-ray is used for follow-up in patients with radiopaque stones, while a KUB CT scan is used otherwise. The primary outcome measure is the stone-free rate after two and twelve weeks, considered as the absence of a stone ≥ 4 mm. Secondary outcome measures include pain after 24 hours, need for re-ESWL, and need for surgery.

Before statistical analysis, adjudication of all measurements will be done by an experienced statistician outside of the research group. The adjudicator will assess the quality of each measurement and will exclude those with inadequate quality from the analysis, where they will be regarded as missing. Once the adjudication process is complete, the finalized database will be unblinded.

Data will be kept anonymous until analysis, which is to be performed by an independent statistician external to the research group. Data are analyzed using SPSS version 25 (IBM, Armonk, NY, USA). Quantitative variables will be compared using the independent t-test or Mann-Whitney U test as appropriate. Qualitative variables will be compared with the chi-squared test or Fisher's exact test as appropriate. Logistic regression will be used to compare the likelihood of success between the study groups after controlling for study variables. P-values below 0.05 indicate statistical significance in all cases.

The study's executive committee will report any adverse events to an independent Data and Safety and Monitoring Board (DSMB). The DSMB will halt the trial if patient safety is compromised or if the primary research objective is met. The DSMB will monitor all safety issues, and the DSMB statistician will report safety problems in each study group monthly. Any deaths will be investigated.

The Ethics Committee of Shiraz University of Medical Sciences approved the study protocol (code: IR.SUMS.MED.REC.1399.085). Informed consent will be obtained from all patients while they are clinically stable and not under the influence of sedatives. All participants are able to withdraw from the study at any point. Given that furosemide does not adversely affect patients who do not have cardiovascular or renal diseases, no complications were predicted. The principles of the Declaration of Helsinki will be upheld throughout this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* Patients with renal or ureteral calculi referred by attending urologists to the ESWL Clinic of Shahid Faghihi Hospital, affiliated to Shiraz University of Medical Sciences (Shiraz, Iran)

Exclusion Criteria:

* An anatomic anomaly in urinary system
* Coagulopathy
* Untreated urinary tract infection
* Prior urologic surgery
* Simultaneous unilateral renal and ureteral stones
* Kidney failure (serum creatinine > 1.8 mg/dl)
* Cardiovascular disease
* Hypertension
* Morbid obesity (BMI > 40 kg/m2)
* History of allergy to furosemide, glibenclamide, hydrochlorothiazide, or acetazolamide.
* Pregnancy
* Single kidney

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate | 2 weeks after intervention
  The absence of a stone ≥ 4 mm
Stone-free rate | 3 months after intervention
  The absence of a stone ≥ 4 mm

SECONDARY OUTCOMES:
Renal colic on VAS of 0-10 | 24 hours after intervention
  Pain related to ureteral or renal calculi within 24 hours of ESWL
Number of participants with need for re-ESWL | Within 3 months after intervention
  The need for a repeated ESWL procedure
Number of participants with need for surgery | Within 3 months after intervention
  The need for a surgery to remove the stone

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Irani, MD, Study Director — Department of Urology, School of Medicine, Shiraz University of Medical Sciences
Locations (1):
- Shahid Faghihi Hospital, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Yes
Yes We plan to publish the study protocol soon. The final results will be published in the form of an article after the study is completed.
Supporting Information: Study Protocol
Time Frame: We plan to publish the study protocol within six months.
Access Criteria: Supporting data will be made available upon reasonable request. All inquiries should be sent to Dr. Seyed Hossein Hosseini.

REFERENCES:
- [Background] Liu Y, Chen Y, Liao B, Luo D, Wang K, Li H, Zeng G. Epidemiology of urolithiasis in Asia. Asian J Urol. 2018 Oct;5(4):205-214. doi: 10.1016/j.ajur.2018.08.007. Epub 2018 Sep 6. PMID 30364478
- [Background] Safarinejad MR. Adult urolithiasis in a population-based study in Iran: prevalence, incidence, and associated risk factors. Urol Res. 2007 Apr;35(2):73-82. doi: 10.1007/s00240-007-0084-6. Epub 2007 Mar 15. PMID 17361397
- [Background] Ketabchi AA, Aziziolahi GA. Prevalence of symptomatic urinary calculi in Kerman, Iran. Urol J. 2008 Summer;5(3):156-60. PMID 18825621
- [Background] Basiri A, Shakhssalim N, Khoshdel AR, Ghahestani SM, Basiri H. The demographic profile of urolithiasis in Iran: a nationwide epidemiologic study. Int Urol Nephrol. 2010 Mar;42(1):119-26. doi: 10.1007/s11255-009-9588-z. Epub 2009 Jun 12. PMID 19521794
- [Background] Sabharwal S, Jeyaseelan L, Panda A, Gnanaraj L, Kekre NS, Devasia A. A prospective randomised double-blind placebo-controlled trial to assess the effect of diuretics on shockwave lithotripsy of calculi. Arab J Urol. 2017 Jul 8;15(4):289-293. doi: 10.1016/j.aju.2017.04.003. eCollection 2017 Dec. PMID 29234530
- [Background] Hosseini MM, Shakeri S, Manaheji F, Aminsharifi A, Ezatzadegan S, Pakfetrat M, Basiratnia M, Hosseini M. Stone composition in patients who undergo renal stone surgery: review of 423 stone analyses in southern iran. Iran J Med Sci. 2014 Jan;39(1):75-6. No abstract available. PMID 24453399
- [Background] McAdams S, Shukla AR. Pediatric extracorporeal shock wave lithotripsy: Predicting successful outcomes. Indian J Urol. 2010 Oct;26(4):544-8. doi: 10.4103/0970-1591.74457. PMID 21369388
- [Background] Azm TA, Higazy H. Effect of diuresis on extracorporeal shockwave lithotripsy treatment of ureteric calculi. Scand J Urol Nephrol. 2002;36(3):209-12. doi: 10.1080/003655902320131893. PMID 12201937
- [Background] Zomorrodi A, Golivandan J, Samady J. Effect of diuretics on ureteral stone therapy with extracorporeal shock wave lithotripsy. Saudi J Kidney Dis Transpl. 2008 May;19(3):397-400. PMID 18445899
- [Background] Sohu S, Soomro MH, Mangrio RH, Shaikh AA, Mirani A, Chand K, Jalbani MH. Efficacy of extracorporeal shockwave lithotripsy with furosemide and hydration in renal stone management: A randomised controlled trial. Arab J Urol. 2019 Jul 24;17(4):279-284. doi: 10.1080/2090598X.2019.1645262. eCollection 2019. PMID 31723445